CLINICAL TRIAL: NCT06581263
Title: Investigating the Use of Virtual Reality in Psychedelic Research or Clinical Practice
Brief Title: Psychedelic Virtual Reality
Status: Recruiting | Type: Observational
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, Anahita Bassir Nia, Assistant Professor of Psychiatry, Yale University
Other Study IDs: 2000038121
Record Dates: First submitted 2024-08-27; First posted 2024-09-03 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Psychedelic Experiences; Virtual Reality; Healthy Volunteer

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy Volunteer
  Interventions: Device: Meta Quest 3

INTERVENTIONS:
Device: Meta Quest 3 — Meta Quest 3 is a virtual reality headset device

SUMMARY:
The purpose of this study is to evaluate a novel VRP.

DETAILED DESCRIPTION:
The primary objective of this study is to determine whether the subjective experience of a novel VRP (DeepDream) will be comparable to a standard dose of psychedelics. This study also looks to compare the subjective experience of DeepDream VRP to other available VR modalities developed to mimic psychedelic subjective experience along with assessing the incidence of VRP adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent
* No history or current DSM-V diagnosis

Exclusion Criteria:

* Unstable medical conditions

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2025-07-22 (Actual); Primary Completion 2026-03-22 (Estimated); Study Completion 2026-03-22 (Estimated)

PRIMARY OUTCOMES:
Assess subjective experience of novel VRP (DeepDream) comparable to a standard dose of psychedelics. | Day 0 through Day 30
  Subject experience will be assessed using the Altered States of Consciousness Rating Scale.
Assess subjective experience of novel VRP (DeepDream) comparable to a standard dose of psychedelics. | Day 0 through Day 30
  Subject experience will be assessed using the Mystical Experience Questionnaire.
Assess subjective experience of novel VRP (DeepDream) comparable to a standard dose of psychedelics. | Day 0 through Day 30
  Subject experience will be assessed using the Ego-Dissolution Inventory.

SECONDARY OUTCOMES:
Assess the incidence of VRP adverse effects, principally virtual reality sickness (VRS) and neck and upper back pain. | Day 0 through Day 30
  The number of adverse events will be assessed through qualitative interviews following VRP viewing.

CONTACTS AND LOCATIONS:
Overall Officials: Anahita Bassir Nia, MD, Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States